CLINICAL TRIAL: NCT04410328
Title: A Randomized Controlled Trial to Evaluate the Outcomes With Aggrenox in Patients With SARS-CoV-2 Infection
Brief Title: Aggrenox To Treat Acute Covid-19
Acronym: ATTAC-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Amit Singla, MD, FAANS, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2020001469
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Covid19
Keywords: COVID-19; SARS-CoV; Aggrenox; Dipyridamole; Aspirin
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Aspirin; Standard of Care; Aspirin, Dipyridamole Drug Combination

STUDY DESIGN:
Intervention Model Description: Arm 1: Aggrenox plus standard care. Participants will receive Aggrenox (Dipyridamole ER 200mg/ Aspirin 25mg orally/enterally), 2 times daily (FDA-recommended dose) starting on the day of enrollment for a total of 2 weeks.
  Arm 2: Standard care. Participants will receive standard care starting on the day of enrollment for a total of 2 weeks.
  The investigators will perform a randomized, 2-arm, open-label single-site pilot study to evaluate the effect of oral Aggrenox (Dipyridamole ER 200mg/ Aspirin 25mg orally/enterally), on clinical outcomes in patients with SARS-CoV-2. In this research proposal, the investigators will randomly assign 132 consenting participants with diagnosis of SARS-CoV-2 to two treatment groups: 1) Aggrenox (Dipyridamole ER 200mg/ Aspirin 25mg orally/enterally) + standard care and 2) standard care alone. Participants will be screened, enrolled, receive treatment and followed for 28 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Participants receiving Dipyridamole and Aspirin (Experimental): Dipyridamole ER 200mg/ Aspirin 25mg orally/enterally plus standard care. Participants will receive Dipyridamole ER 200mg/ Aspirin 25mg orally/enterally), 2 times daily starting on the day of enrollment for a total of 2 weeks.
  Interventions: Drug: Dipyridamole ER 200mg/ Aspirin 25mg orally/enterally AND Standard of care; Other: Standard of care
- Participants receiving standard of care (Other): Participants will receive standard care starting on the day of enrollment for a total of 2 weeks. Standard of care treatment consist of an intravenous Remidesivir 200 mg loading dose and then 100 mg/daily for a total of 4 days for non-intubated patients and 10 days for intubated patients, intravenous/oral decadron 6 mg/daily for 10 days and prophylactic subcutaneous LMWH daily, started on the day of enrollment and for the duration of hospitalization. If the patients are discharged before 10 days, they are prescribed oral decadron 6 mg daily to complete the course of 10 days.
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: Dipyridamole ER 200mg/ Aspirin 25mg orally/enterally AND Standard of care — Participants in the experimental group will receive Dipyridamole ER 200mg/ Aspirin 25mg orally/enterally (if they have a feeding tube), 2 times daily starting on the day of enrollment for a total of 2 weeks.
  Other Names: Aggrenox
  Arms: Participants receiving Dipyridamole and Aspirin
Other: Standard of care — Participants will receive standard care starting on the day of enrollment for a total of 2 weeks. Standard of care treatment consist of an intravenous Remidesivir 200 mg loading dose and then 100 mg/daily for a total of 4 days for non-intubated patients and 10 days for intubated patients, intravenous/oral decadron 6 mg/daily for 10 days and prophylactic subcutaneous LMWH daily, started on the day of enrollment and for the duration of hospitalization. If the patients are discharged before 10 days, they are prescribed oral decadron 6 mg daily to complete the course of 10 days.

SUMMARY:
The purpose of this study is to explore the efficacy of Aggrenox in patients with SARS-CoV-2 infection with symptoms consistent with COVID-19. An anticipated total of 132 participants will be randomly divided almost equally into 2 groups: one group will receive Dipyridamole ER 200mg/ Aspirin 25mg orally/enterally along with the standard of care and the other group with receive the standard of care only but no Dipyridamole ER 200mg/ Aspirin 25mg. Participants will be screened, enrolled, receive treatment, and followed for 28 days. The clinical and laboratory outcomes of all the participants enrolled in the study will be evaluated at the end of the study to explore if there is any difference in the outcomes between 2 groups.

DETAILED DESCRIPTION:
Purpose/Specific Aims: The purpose of this study is to explore the efficacy of Aggrenox in patients with SARS-CoV-2 infection with symptoms consistent with COVID-19.

Among 132 SARS-CoV-2 patients (66 patients in each randomized arm), we will determine the efficacy of Aggrenox on clinical outcomes.

Hypotheses / Research Question(s) Compared to standard care, the addition of Aggrenox (Dipyridamole ER 200mg/ Aspirin 25mg), to standard care will result in improvement in the composite COVID ordinal scale at day 15. Additionally, combined Aggrenox (Dipyridamole ER 200mg/ Aspirin 25mg orally/enterally), and standard care will reduce the need for ventilation, length of mechanical ventilation, hospital length of stay, ICU length of stay, decrease risk of thromboembolic complications and improve survival more than standard care alone in SARS-CoV-2 patients.

Research Design and Methods Randomized design. Participants will be randomized 1:1 to Aggrenox or standard treatment. Arm 1: Active Comparator: (Aggrenox (Dipyridamole ER 200mg/ Aspirin 25mg orally/enterally).

Participants will receive Aggrenox (Dipyridamole ER 200mg/ Aspirin 25mg orally/enterally), 2 times daily (FDA-recommended dose) starting on the day of enrollment for a total of 2 weeks + standard care.

Arm 2: Standard care Comparator: Participants will receive standard care starting on the day of enrollment for a total of 2 weeks.

The investigators will perform a randomized, 2-arm, open-label single-site pilot study to evaluate the effect of oral Aggrenox (Dipyridamole ER 200mg/ Aspirin 25mg orally/enterally), on clinical outcomes in patients with SARS-CoV-2. In this research proposal, investigators will randomly assign 132 consenting participants with diagnosis of SARS-CoV-2 to two treatment groups: 1) Aggrenox (Dipyridamole ER 200mg/ Aspirin 25mg orally/enterally) + standard care and 2) standard care alone. Participants will be screened, enrolled, receive treatment and followed for 28 days. The study aim and procedure will be explained to every eligible subject and informed consent will be obtained from interested subjects or authorized proxy to participate in the study. The investigators will collect demographic, clinical, laboratory and radiological data. The patients would be followed daily for 2 weeks after enrollment while the patient is in the hospital and once discharged, they will be called every 3rd day to follow up on the symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Hospitalization.
3. SARS-CoV-2 viral nucleic acid positive within 3 days.
4. Lab test result pending plus a high clinical suspicion for SARS-CoV-2 (fever and cough for ≤ 7 days, bilateral pulmonary infiltrates on imaging or new hypoxemia with spO2 ≤94% on room air or no alternative explanation for respiratory symptoms).
5. Willing and able to provide consent or by authorized proxy.

Exclusion Criteria:

1. Pregnancy.
2. G-6PD deficiency.
3. Use of antiplatelet agents including inhibitor of P2Y12 ADP platelet receptors, phosphodiesterase inhibitors, and Glycoprotein IIB/IIIA inhibitors.
4. On therapeutic anticoagulation with coumadin, heparin and direct oral anticoagulants.
5. Vasodilatory shock.
6. Patient with known ongoing angina, recent myocardial infarction and sub-valvular aortic stenosis.
7. Active gastric or duodenal ulcer or any bleeding disorder.
8. Hemoglobin <9 mg/dL, platelet count of <30,000 /mm3.
9. Acute respiratory infection for >10 days.
10. Known allergy/hypersensitivity to Dipyridamole and/or Aspirin.
11. Severe hepatic or renal insufficiency.
12. Uncontrolled hypertension defined as systolic > 180 mm Hg or diastolic > 100 mm Hg.
13. Patients with known allergy to NSAIDs

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Singla, MD, Principal Investigator — Rutgers University
Locations (1):
- Rutgers New Jersey Medical School University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Macatangay BJC, Jackson EK, Abebe KZ, Comer D, Cyktor J, Klamar-Blain C, Borowski L, Gillespie DG, Mellors JW, Rinaldo CR, Riddler SA. A Randomized, Placebo-Controlled, Pilot Clinical Trial of Dipyridamole to Decrease Human Immunodeficiency Virus-Associated Chronic Inflammation. J Infect Dis. 2020 Apr 27;221(10):1598-1606. doi: 10.1093/infdis/jiz344. PMID 31282542
- [Result] Li Z LX, Huang Yi-Y et al. FEP-based screening prompts drug repositioning against COVID-19. 2020.
- [Result] Liu X LZ, Liu S et al. . Therapeutic effects of dipyridamole on COVID-19 patients with coagulation dysfunction. 2020.
- [Result] Kohler D, Streienberger A, Morote-Garcia JC, Granja TF, Schneider M, Straub A, Boison D, Rosenberger P. Inhibition of Adenosine Kinase Attenuates Acute Lung Injury. Crit Care Med. 2016 Apr;44(4):e181-9. doi: 10.1097/CCM.0000000000001370. PMID 26491864
- [Result] Fata-Hartley CL, Palmenberg AC. Dipyridamole reversibly inhibits mengovirus RNA replication. J Virol. 2005 Sep;79(17):11062-70. doi: 10.1128/JVI.79.17.11062-11070.2005. PMID 16103157
- [Result] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Receiving Dipyridamole and Aspirin: Dipyridamole ER 200mg/ Aspirin 25mg orally/enterally plus standard care. Participants will receive Dipyridamole ER 200mg/ Aspirin 25mg orally/enterally), 2 times daily starting on the day of enrollment for a total of 2 weeks.
  Dipyridamole ER 200mg/ Aspirin 25mg orally/enterally AND Standard of care: Participants in the experimental group will receive Dipyridamole ER 200mg/ Aspirin 25mg orally/enterally (if they have a feeding tube), 2 times daily starting on the day of enrollment for a total of 2 weeks.
  Standard of care: Participants will receive standard care starting on the day of enrollment for a total of 2 weeks.
- Participants Receiving Standard of Care: Participants will receive standard care starting on the day of enrollment for a total of 2 weeks.
  Standard of care: Participants will receive standard care starting on the day of enrollment for a total of 2 weeks.
  Standard of care treatment consist of an intravenous Remidesivir 200 mg loading dose and then 100 mg/daily for a total of 4 days for non-intubated patients and 10 days for intubated patients, intravenous/oral decadron 6 mg/daily for 10 days and prophylactic subcutaneous LMWH daily, started on the day of enrollment and for the duration of hospitalization. If the patients are discharged before 10 days, they are prescribed oral decadron 6 mg daily to complete the course of 10 days
Period: Overall Study
Arm/Group | Participants Receiving Dipyridamole and Aspirin | Participants Receiving Standard of Care
Started | 49 | 49
Completed | 49 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants Receiving Standard of Care: Participants will receive standard care starting on the day of enrollment for a total of 2 weeks.
  Standard of care: Participants will receive standard care starting on the day of enrollment for a total of 2 weeks.
- Total: Total of all reporting groups
Arm/Group | Participants Receiving Dipyridamole and Aspirin | Participants Receiving Standard of Care | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 49 | 98
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57.5 [47 to 63] | 56 [47 to 62] | 57 [47 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 21 | 52
  Male | 18 | 28 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 9 | 9 | 18
  East Asian | 0 | 0 | 0
  South Asian | 0 | 1 | 1
  West Asian | 0 | 0 | 0
  Latin American | 10 | 10 | 20
  White | 1 | 0 | 1
  Aboriginal/First Nations | 0 | 0 | 0
  Mixed | 0 | 1 | 1
  Other | 2 | 3 | 5
  Unknown | 27 | 25 | 52
Region of Enrollment [Number; unit: participants]
  United States | 49 | 49 | 98

OUTCOME MEASURES:

1. Primary Outcome: Covid (Coronavirus Disease-19) Ordinal Scale
Description: Change in composite COVID ordinal scale from day 1 to 14. Ordinal scale: 1) not hospitalized with resumption of normal activities; 2) not hospitalized, but unable to resume normal activities; 3) hospitalized, not requiring oxygen; 4) hospitalized, requiring oxygen; 5) hospitalized, requiring high-flow oxygen therapy, or noninvasive ventilation; 6) hospitalized, requiring invasive ventilation; 7) ventilation plus additional organ support such as pressors, renal replacement therapy and ECMO and 8) death.
  COVID Ordinal Scale ranges from 1 to 8, with score 1 on the scale corresponds to an ambulatory patient with minimal symptoms and score 8 on the scale corresponds to death.
Time Frame: 15 days
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Participants Receiving Dipyridamole and Aspirin | Participants Receiving Standard of Care
Number analyzed (Participants) | 49 | 49
score on a scale | 2.3 (1.8) | 2.1 (2.0)

2. Secondary Outcome: Mortality
Description: All-cause mortality assessed on day 14.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Dipyridamole and Aspirin | Participants Receiving Standard of Care
Number analyzed (Participants) | 49 | 49
Participants | 2 | 2

3. Secondary Outcome: Mortality
Description: All-cause mortality assessed on day 28.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Dipyridamole and Aspirin | Participants Receiving Standard of Care
Number analyzed (Participants) | 49 | 49
Participants | 3 | 5

4. Secondary Outcome: Inflammatory Marker Between Baseline and 7 Days
Description: Change in marker D-dimer
Time Frame: Baseline and 7 days
Measure: Median (Inter-Quartile Range); unit: ng/mL
Groups:
- Participants Receiving Dipyridamole and Aspirin: Dipyridamole ER 200mg/ Aspirin 25mg orally/enterally AND Standard of care: Participants in the experimental group will receive Dipyridamole ER 200mg/ Aspirin 25mg orally/enterally (if they have a feeding tube), 2 times daily starting on the day of enrollment for a total of 2 weeks.
  Standard of care: Participants will receive standard care starting on the day of enrollment for a total of 2 weeks.
Arm/Group | Participants Receiving Dipyridamole and Aspirin | Participants Receiving Standard of Care
Number analyzed (Participants) | 49 | 49
ng/mL | -197.5 [-2425.0 to 366.0] | 114 [-1408.0 to 240.0]

5. Secondary Outcome: COVID Ordinal Scale
Description: COVID ordinal scale
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Participants Receiving Dipyridamole and Aspirin | Participants Receiving Standard of Care
Number analyzed (Participants) | 49 | 49
scores on a scale | 3 [2 to 4] | 3 [2 to 3]

6. Secondary Outcome: Number of Participants Not Requiring Supplemental Oxygen
Description: number of participants who received supplemental oxygen or those with supplemental oxygen-free days
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Dipyridamole and Aspirin | Participants Receiving Standard of Care
Number analyzed (Participants) | 49 | 49
Participants | 45 | 43

7. Secondary Outcome: Invasive-ventilator
Description: Number of participants who were invasive-ventilator free
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Dipyridamole and Aspirin | Participants Receiving Standard of Care
Number analyzed (Participants) | 49 | 49
Participants | 4 | 5

8. Secondary Outcome: ICU Stay
Description: Number of participants admitted to ICU
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Dipyridamole and Aspirin | Participants Receiving Standard of Care
Number analyzed (Participants) | 49 | 49
Participants | 5 | 7

9. Secondary Outcome: Inflammatory Marker
Description: Increase in marker Ferritin
Time Frame: Baseline and 7 days
Measure: Median (Inter-Quartile Range); unit: ug/L
Arm/Group | Participants Receiving Dipyridamole and Aspirin | Participants Receiving Standard of Care
Number analyzed (Participants) | 49 | 49
ug/L | 652.5 [312 to 1752] | 381 [115 to 521]

10. Secondary Outcome: Inflammatory Marker
Description: Increase in marker C-reactive protein
Time Frame: Baseline and 7 days
Measure: Median (Inter-Quartile Range); unit: ug/L
Arm/Group | Participants Receiving Dipyridamole and Aspirin | Participants Receiving Standard of Care
Number analyzed (Participants) | 49 | 49
ug/L | 92 [83 to 101] | 165 [85 to 262]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a period of 28 days.
Description: Study participants death was a result of their diagnosis and not due to the study intervention.
Arm/Group | Participants Receiving Dipyridamole and Aspirin | Participants Receiving Standard of Care
All-Cause Mortality (participants affected / at risk) | 5/49 | 7/49
Serious Adverse Events (participants affected / at risk) | 5/49 | 7/49
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Receiving Dipyridamole and Aspirin (N=49) | Participants Receiving Standard of Care (N=49)
death (Infections and infestations) | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT04410328/Prot_SAP_003.pdf
  • Informed Consent Form (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT04410328/ICF_004.pdf